CLINICAL TRIAL: NCT01377233
Title: A Randomised, Double-blind, Parallel-group, Explorative Study of the Safety, Tolerability, and Pharmacokinetics of Daily Dosing Compared to Weekly Dosing of Zicronapine in Patients With Schizophrenia
Brief Title: Study of the Safety, Tolerability, and Pharmacokinetics of Once Weekly Zicronapine in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13946A
Record Dates: First submitted 2011-06-20; First posted 2011-06-21 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic; Zicronapine; Lu 31-310
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Zicronapine open-label lead-in 10 mg daily (Experimental)
  Interventions: Drug: Zicronapine open-label lead-in 10 mg daily
- Zicronapine 10 mg daily (Experimental)
  Interventions: Drug: Zicronapine 10 mg daily
- Zicronapine 20 mg once weekly (Experimental)
  Interventions: Drug: Zicronapine 20 mg once weekly
- Zicronapine 30 mg once weekly (Experimental)
  Interventions: Drug: Zicronapine 30 mg once weekly
- Zicronapine 45 mg once weekly (Experimental)
  Interventions: Drug: Zicronapine 45 mg once weekly

INTERVENTIONS:
Drug: Zicronapine open-label lead-in 10 mg daily — Encapsulated tablet ,10 mg, once daily, open-label
  Other Names: Lu 31-130
  Arms: Zicronapine open-label lead-in 10 mg daily
Drug: Zicronapine 10 mg daily — Encapsulated tablet, 10 mg, once daily, double-blind
  Other Names: Lu 31-130
  Arms: Zicronapine 10 mg daily
Drug: Zicronapine 20 mg once weekly — Encapsulated tablet, 20 mg, once weekly (on day 1 of each 7 day cycle), double-blind
  Other Names: Lu 31-130
  Arms: Zicronapine 20 mg once weekly
Drug: Zicronapine 30 mg once weekly — Encapsulated tablet, 30 mg, once weekly (on day 1 of each 7 day cycle), double-blind
  Other Names: Lu 31-130
  Arms: Zicronapine 30 mg once weekly
Drug: Zicronapine 45 mg once weekly — Encapsulated tablet, 45 mg, once weekly (on day 1 of each 7 day cycle), double-blind
  Other Names: Lu 31-130
  Arms: Zicronapine 45 mg once weekly

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of once weekly dosing of zicronapine, compared to daily dosing of zicronapine.

DETAILED DESCRIPTION:
The study includes 2 treatment periods. The open-label run-in period will begin at patient enrolment and continue for 3 weeks, during which all patients will receive once daily treatment with zicronapine. The double-blind period will begin at patient randomization and continue for 5 weeks, during which the patients will be assigned to one group receiving once daily treatment with zicronapine and 3 groups receiving once weekly treatment with zicronapine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR)
* A score of <=4 (moderately ill) on Clinical Global Impression - Severity of Illness (CGI-S) scale
* A total score >=60 on Positive and Negative Syndrome Scale (PANSS)
* A score of <=4 (moderate) on PANSS items: P7 (hostility) AND G8 (uncooperativeness)

Exclusion Criteria:

* Acute exacerbation requiring hospitalization within the last 3 months OR requiring change of antipsychotic medication within the last 4 weeks
* Diagnosis or history of substance dependence or substance abuse according to DSM-IV-TR within the last 3 months
* Significant risk of harming himself/herself or others
* Positive serology for hepatitis A, B, C, or HIV
* Present condition that might compromise liver function
* Medical or neurological disorder or treatment that could interfere with study treatment or compliance
* Previous exposure to zicronapine

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (4):
- United States (4):
  - US002, Garden Grove, California
  - US003, National City, California
  - US004, San Diego, California
  - US001, Rockville, Maryland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 46 patients were initially enrolled in a 3-week open-label study period. The 42 patients who completed the open-label period were subsequently randomized to a 5-week double-blind period.
Groups:
- Zicronapine Open-label 10 mg Daily: Zicronapine open-label 10 mg daily: Encapsulated tablet ,10 mg, once daily, open-label
- Zicronapine Basis Dose 10 mg Daily: Zicronapine basis dose 10 mg daily: Encapsulated tablet, 10 mg, once daily, double-blind
- Zicronapine Low Dose 20 mg Once Weekly: Zicronapine low dose 20 mg once weekly: Encapsulated tablet, 20 mg, once weekly (on day 1 of each 7 day cycle), double-blind
- Zicronapine Med Dose 30 mg Once Weekly: Zicronapine med dose 30 mg once weekly: Encapsulated tablet, 30 mg, once weekly (on day 1 of each 7 day cycle), double-blind
- Zicronapine High Dose 45 mg Once Weekly: Zicronapine high dose 45 mg once weekly: Encapsulated tablet, 45 mg, once weekly (on day 1 of each 7 day cycle), double-blind
Period: Open-label
Arm/Group | Zicronapine Open-label 10 mg Daily | Zicronapine Basis Dose 10 mg Daily | Zicronapine Low Dose 20 mg Once Weekly | Zicronapine Med Dose 30 mg Once Weekly | Zicronapine High Dose 45 mg Once Weekly
Started | 46 | 0 | 0 | 0 | 0
Completed | 42 | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0 | 0
Period: Double-blind
Arm/Group | Zicronapine Open-label 10 mg Daily | Zicronapine Basis Dose 10 mg Daily | Zicronapine Low Dose 20 mg Once Weekly | Zicronapine Med Dose 30 mg Once Weekly | Zicronapine High Dose 45 mg Once Weekly
Started | 0 | 11 | 10 | 11 | 10
Completed | 0 | 10 | 8 | 7 | 8
Not Completed | 0 | 1 | 2 | 4 | 2
Not completed — Adverse Event | 0 | 1 | 2 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Administrative or other | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for the 4 patients enrolled in the open-label period but not randomized to the double blinded period, are reported in the first (open-label) study arm. Baseline characteristics for the 42 patients who were subsequently randomized to the double-blind period are reported across the last four (randomized) study arms.
Groups:
- Zicronapine 10 mg Daily: Zicronapine basis dose 10 mg daily: Encapsulated tablet, 10 mg, once daily, double-blind
- Zicronapine 20 mg Once Weekly: Zicronapine low dose 20 mg once weekly: Encapsulated tablet, 20 mg, once weekly (on day 1 of each 7 day cycle), double-blind
- Zicronapine 30 mg Once Weekly: Zicronapine med dose 30 mg once weekly: Encapsulated tablet, 30 mg, once weekly (on day 1 of each 7 day cycle), double-blind
- Zicronapine 45 mg Once Weekly: Zicronapine high dose 45 mg once weekly: Encapsulated tablet, 45 mg, once weekly (on day 1 of each 7 day cycle), double-blind
- Total: Total of all reporting groups
Arm/Group | Zicronapine Open-label 10 mg Daily | Zicronapine 10 mg Daily | Zicronapine 20 mg Once Weekly | Zicronapine 30 mg Once Weekly | Zicronapine 45 mg Once Weekly | Total
Number analyzed (Participants) | 4 | 11 | 10 | 11 | 10 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (6.6) | 42.7 (11.7) | 47.8 (6.4) | 50.8 (5.0) | 50.1 (4.8) | 47.0 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 4 | 4 | 4 | 17
  Male | 3 | 7 | 6 | 7 | 6 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 7 | 5 | 8 | 7 | 28
  White | 2 | 4 | 4 | 3 | 3 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 11 | 10 | 11 | 10 | 46
Height [Mean (Standard Deviation); unit: cm] | 176.3 (9.4) | 169.5 (8.3) | 170.1 (9.7) | 174.6 (10.3) | 170.9 (11.7) | 171.8 (9.8)
Weight [Mean (Standard Deviation); unit: kg] | 94.7 (27.5) | 90.0 (21.1) | 91.5 (19.2) | 87.5 (17.5) | 93.8 (16.8) | 89.7 (18.0)
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.0 (5.5) | 31.3 (7.1) | 31.6 (5.9) | 28.6 (4.2) | 32.2 (5.2) | 30.4 (5.3)
Waist circumference [Mean (Standard Deviation); unit: cm] | 98.7 (16.2) | 99.8 (16.4) | 101.8 (14.1) | 101.1 (13.1) | 106.5 (12.5) | 103.3 (13.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events as a Measure of Safety and Tolerability
Description: Number of patients with treatment-emergent adverse events during each of the two study periods plus corresponding safety follow-up period. Open-label period: 3 weeks post-baseline plus 8 weeks safety follow-up (11 weeks total); Double-blind period: 5 weeks post-randomization plus 8 weeks safety follow-up (13 weeks total)
Time Frame: 11 weeks for open-label period; 13 weeks for double-blind period
Population: Adverse events for the 46 patients enrolled in the open-label period are reported in the first (open-label) study arm. Adverse events for the 42 patients (out of the 46 enrolled) who were subsequently randomized to the double-blind period are reported across the last four (randomized) study arms.
Measure: Number; unit: participants
Arm/Group | Zicronapine Open-label 10 mg Daily | Zicronapine Basis Dose 10 mg Daily | Zicronapine Low Dose 20 mg Once Weekly | Zicronapine Med Dose 30 mg Once Weekly | Zicronapine High Dose 45 mg Once Weekly
Number analyzed (Participants) | 46 | 11 | 10 | 11 | 10
participants | 12 | 8 | 4 | 4 | 9

2. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) Total and Subscales Change From Baseline
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 that indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. The PANSS total score was the sum of the rating scores for 7 positive subscale items, 7 negative subscale items, and 16 general psychopathology subscale items from the PANSS panel. PANSS Total Score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: 8 weeks post-baseline (3 weeks open-label period plus 5 weeks double-blind period)
Population: All patients who were randomized to the double-blind study period, who took at least one dose of drug, and who had at least one valid PANSS assessment were included in the analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zicronapine Basis Dose 10 mg Daily | Zicronapine Low Dose 20 mg Once Weekly | Zicronapine Med Dose 30 mg Once Weekly | Zicronapine High Dose 45 mg Once Weekly
Number analyzed (Participants) | 10 | 8 | 7 | 8
units on a scale
  PANSS total | -8.0 (2.7) | -8.7 (2.5) | -10.6 (2.6) | -12.2 (2.5)
  PANSS Positive Symptoms | -1.5 (1.1) | -0.8 (1.0) | -1.8 (1.1) | -2.6 (1.0)
  PANSS Negative Symptoms | -2.9 (1.0) | -2.8 (1.0) | -2.0 (1.0) | -3.1 (1.0)
  PANSS General Psychopathology | -5.2 (1.2) | -5.5 (1.2) | -6.4 (1.3) | -6.2 (1.2)

3. Secondary Outcome: Clinical Global Impression Severity Scale (CGI-S) Change From Baseline
Description: The CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses their clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients).
Time Frame: 8 weeks post-baseline (3 weeks open-label period plus 5 weeks double-blind period)
Population: All patients who were randomized to the double-blind study period, who took at least one dose of drug, and who had at least one valid PANSS assessment were included in the full analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Zicronapine Basis Dose 10 mg Daily | Zicronapine Low Dose 20 mg Once Weekly | Zicronapine Med Dose 30 mg Once Weekly | Zicronapine High Dose 45 mg Once Weekly
Number analyzed (Participants) | 10 | 8 | 7 | 8
units on a scale | -0.5 (0.2) | -0.5 (0.2) | -0.2 (0.2) | -0.7 (0.2)

4. Secondary Outcome: Clinical Global Impression Improvement Scale (CGI-I)
Description: The CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). In all cases, the assessment is made independent of whether the rater believes the improvement is drug-related or not.
Time Frame: 8 weeks post-baseline (3 weeks open-label period plus 5 weeks double-blind period)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zicronapine Basis Dose 10 mg Daily | Zicronapine Low Dose 20 mg Once Weekly | Zicronapine Med Dose 30 mg Once Weekly | Zicronapine High Dose 45 mg Once Weekly
Number analyzed (Participants) | 10 | 8 | 7 | 8
units on a scale | 2.9 (0.6) | 3.4 (1.1) | 3.0 (0.6) | 2.9 (1.1)

ADVERSE EVENTS:
Time Frame: Open-label period: 3 weeks post-baseline plus 8 weeks safety follow-up (11 weeks total); Double-blind period: 5 weeks post-randomization plus 8 weeks safety follow-up (13 weeks total)
Description: Adverse events were monitored at all study visits incl. screening, baseline, completion/withdrawal and safety follow-up visits. All adverse events observed by investigators or reported by patients were recorded. Results from relevant clinical safety tests were also recorded as adverse events if considered clinically significant by the investigator.
Arm/Group | Zicronapine Open-label 10 mg Daily | Zicronapine Basis Dose 10 mg Daily | Zicronapine Low Dose 20 mg Once Weekly | Zicronapine Med Dose 30 mg Once Weekly | Zicronapine High Dose 45 mg Once Weekly
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/11 | 1/10 | 1/11 | 1/10
Other Adverse Events (participants affected / at risk) | 8/46 | 8/11 | 4/10 | 4/11 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zicronapine Open-label 10 mg Daily (N=46) | Zicronapine Basis Dose 10 mg Daily (N=11) | Zicronapine Low Dose 20 mg Once Weekly (N=10) | Zicronapine Med Dose 30 mg Once Weekly (N=11) | Zicronapine High Dose 45 mg Once Weekly (N=10)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zicronapine Open-label 10 mg Daily (N=46) | Zicronapine Basis Dose 10 mg Daily (N=11) | Zicronapine Low Dose 20 mg Once Weekly (N=10) | Zicronapine Med Dose 30 mg Once Weekly (N=11) | Zicronapine High Dose 45 mg Once Weekly (N=10)
Ventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight Increased (Investigations) | 0 | 2 | 1 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Sedation (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
Tardive Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Drug Abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 2 | 0 | 1
Libido Decreased (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Treatment Noncompliance (Social circumstances) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No